CLINICAL TRIAL: NCT04480541
Title: A Pilot Study of Roadmap 2.0 in Oncology Caregivers and Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UMCC 2020.040; HUM00176584 (Other: University of Michigan Rogel Cancer Center)
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Cancer; Quality of Life
Keywords: Mobile Health Technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Roadmap 2.0 + Fitbit Charge 3 (Experimental): * Caregivers and patients download the Roadmap 2.0 mobile app on their own mobile phones or tablet to use freely throughout the 120 day study period.
  * Caregivers and patients receive a Fitbit wearable activitiy sensor to track activity and sleep.
  Interventions: Behavioral: Roadmap 2.0 information system; Other: Wearable activity sensor; Other: Survey administration

INTERVENTIONS:
Behavioral: Roadmap 2.0 information system — Caregivers and patients download the Roadmap 2.0 app on their own mobile phones/tablet
Other: Wearable activity sensor — Caregivers and patients will receive a Fitbit wearable activity sensor
  Other Names: Fitbit Charge 3
Other: Survey administration — Caregivers and patients will be asked to complete health-related quality of life surveys
  Other Names: PROMIS®

SUMMARY:
This study will investigate the use of a mobile health app (Roadmap 2.0) intervention in caregivers of patients with cancer. In this study participants will be given the Roadmap 2.0 app, with a focus on the positive aspects of caregiving (positive activity components), and a Fitbit. The primary objective of this pilot study is to test the feasibility and acceptability of using the mobile health app.

DETAILED DESCRIPTION:
Health information technology tools may enable caregivers and patients to become more active participants in their healthcare.This study is not to provide any treatment, but rather to investigate the use of this mobile health technology-mediated intervention (Roadmap 2.0).

ELIGIBILITY:
Inclusion Criteria:

1. The caregiver must have an eligible patient (defined in items 5 - 9, below)
2. The caregiver must be of age ≥18 years.
3. The caregiver should be comfortable in reading and speaking English and signing informed consents.
4. The caregiver should provide at least 50% of care needs.
5. An eligible patient is one who identifies the eligible caregiver as their primary caregiver (i.e., provides at least 50% of care needs). The caregiver who provides consent will be deemed the caregiver who participates in the study. In adolescents who are at the age to provide assent, she/he will designate the caregiver who provides >50% of their care, and that caregiver will sign the consent document.
6. An eligible patient is age ≥5 years.
7. An eligible patient is able to sign informed consent/assent forms.
8. Patients and caregivers agree to provide informed consent that is in regulatory compliance and IRBMED-approved.
9. The caregiver and patient must have his/her own smartphone or tablet to participate.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Roadmap 2.0 login rate | Day 120
  Percentage of participants (caregivers and patients) who login to Roadmap 2.0 at least 2 times per week for at least 50% of the study duration (120 days). Login data will be collected by the Roadmap 2.0 software. Qualitative and quantitative analysis will be conducted.
Enrollment rate | At time of enrollment
  Percentage of participants (caregivers and patients) enrolled in the study, of the total number approached for enrollment. Qualitative and quantitative analysis will be conducted.

SECONDARY OUTCOMES:
Survey completion rate | Day 120
  Percentage of participants (caregivers and patients) who complete all 3 surveys at each of 3 designated time points: Day 0, day 30 and day 120.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Rogel Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No